CLINICAL TRIAL: NCT01040494
Title: Effects of add-on Aliskiren Treatment on Central and Peripheral Hemodynamics and Biomarkers in Patients With Chronic Congestive Heart Failure (NYHA Class II-IV) (First Year Project)
Brief Title: Add-on Aliskiren Treatment in Patients With Chronic Congestive Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Lian-Yu Lin, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200911004M
Record Dates: First submitted 2009-12-25; First posted 2009-12-29 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-12

CONDITIONS: Congestive Heart Failure
Keywords: Aliskiren; Congestive heart failure; Central hemodynamics
MeSH Terms: conditions — Heart Failure | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren, add-on (Experimental): HF patients will be randomized to receive add-on aliskiren 150 mg for 6 months
  Interventions: Drug: Aliskiren
- placebo, add-on (Placebo Comparator): patients will be randomized to receive add-on placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — all eligible patients will be randomized to receive aliskiren 150 mg on top of optimal HF therapy, including ACEI, ARB, beta blockers as considered appropriate by the investigator and in accordance with standard therapy guidelines for 6 months
  Other Names: rasilez
  Arms: Aliskiren, add-on
Drug: Placebo — all eligible patients will be randomized to receive placebo on top of optimal HF therapy, including ACEI, ARB, beta blockers as considered appropriate by the investigator and in accordance with standard therapy guidelines for 6 months
  Arms: placebo, add-on

SUMMARY:
Aliskiren is a potent direct renin inhibitor and has been recently shown to have favorable neurohumoral effects in patients with heart failure (HF) Objective：To study the effects of add-on aliskiren treatment in patients with HF on components of arterial load, from central aorta to peripheral arterioles and biomarkers Methods：Patients with NYHA Class II to IV HF, who have been treated with angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) and beta-blocker are randomized to 6 months of treatment with placebo or aliskiren (150mg per day) treatment. Components of arterial load, from central aorta to peripheral arterioles as well as a wide-range of biomarkers, including inflammatory biomarkers, N-terminal pro-B type natriuretic peptide, arterial remodeling markers (procollagen, matrix metalloproteinase) will be measured before, 2 months and 6 months after treatment.

What is New or Innovative in this study? The importance of central hemodynamics and biomarker changes in patients with HF has been shown in observation studies. This is the first randomized control trial that examines comprehensively the effects of a direct rennin inhibitor on central hemodynamics and biomarkers in HF patients who are receiving standard heart failure therapy.

DETAILED DESCRIPTION:
Introduction: Aliskiren is a potent direct renin inhibitor and has been recently shown to have favorable neurohumoral effects in patients with heart failure (HF) Objective：To study the effects of add-on aliskiren treatment in patients with HF on components of arterial load, from central aorta to peripheral arterioles and biomarkers Methods：Patients with NYHA Class II to IV HF, who have been treated with angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) and beta-blocker are randomized to 6 months of treatment with placebo or aliskiren (150mg per day) treatment. Components of arterial load, from central aorta to peripheral arterioles as well as a wide-range of biomarkers, including inflammatory biomarkers, N-terminal pro-B type natriuretic peptide, arterial remodeling markers (procollagen, matrix metalloproteinase) will be measured before, 2 months and 6 months after treatment.

What is New or Innovative in this study? The importance of central hemodynamics and biomarker changes in patients with HF has been shown in observation studies. This is the first randomized control trial that examines comprehensively the effects of a direct rennin inhibitor on central hemodynamics and biomarkers in HF patients who are receiving standard heart failure therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients ≥ 18 years of age, male or female. Female patients must be either post-menopausal for one year, surgically sterile, or using effective contraceptive methods such as oral contraceptives, barrier method with spermicide or an intrauterine device.
2. Patients with a diagnosis of chronic heart failure (NYHA Class II-IV) and reduced systolic function: LVEF ≤ 45% at Visit 1 (local measurement, measured within the past 6 months assessed by echocardiogram, MUGA, CT scan, MRI or ventricular angiography).
3. Patients must be on a stable dose of either an ACE inhibitor or an ARB for at least 4 weeks prior to Visit 1.
4. Patients must be treated with a beta blocker, unless contraindicated or not tolerated, at a stable dose for at least 4 weeks prior to Visit 1.
5. Patients with documented sinus rhythm at Visit 1.

Exclusion Criteria:

1. History of hypersensitivity to any of the study drugs.
2. Patients who require treatment with both ACEI and ARB.
3. Current acute decompensated HF (exacerbation of chronic HF manifested by signs & symptoms that may require IV therapy).
4. Symptomatic hypotension and/or less than 100 mmHg at the time of screening or less than 90 mmHg at the time of randomization.
5. eGFR < 30 ml/min/1.73m2 as measured by the MDRD formula at Visit 1 (screening) , or a > 25% decrease after 14 days of active run-in period.
6. Serum potassium > 5.0 mmol/L at screening (Visit 1).
7. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 3 months prior to visit 1.
8. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after Visit 1.
9. Patients with active or unstable bronchospasm or asthma (patients must be on stable regimen of respiratory medications for 1 month prior to Visit 1).
10. Right heart failure due to severe pulmonary disease.
11. Diagnosis of peripartum or chemotherapy induced cardiomyopathy within the 12 months prior to visit 1.
12. Patients with a history of heart transplant or who are on a transplant list or with left ventricular assistance device (LVAD device).
13. Documented ventricular arrhythmia with syncopal episodes within past 3 months, prior to visit 1, that is untreated.
14. Symptomatic bradycardia or second or third degree heart block without a pacemaker.
15. Implantation of a CRT (cardiac resynchronization therapy) device within the prior 3 months from visit 1 or intent to implant a CRT device.
16. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
17. Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis.
18. Severe primary pulmonary, renal or hepatic disease.
19. Presence of any other disease with a life expectancy of < 1 year.
20. Chronic long-term requirement for NSAIDs (high dose) or COX2 inhibitors, with the exception of aspirin at doses used for CV prophylaxis (≤325 mg o.d.).
21. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs
22. Subjects are now breast feeding, get pregnant or will be pregnant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-07 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Central hemodynamics including aortic impedance, central blood pressure, pulse wave velocity | baseline, 2 months, 6 months

SECONDARY OUTCOMES:
Biomarkers including NT-pro-BNP, CRP, MMP | baseline, 2 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lian-Yu Lin, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veteral General Hospital, Taipei